CLINICAL TRIAL: NCT03557918
Title: Phase 2 Trial of Tremelimumab in Patients With Metastatic Urothelial Cancer Previously Treated With PD-1/PD-L1 Blockade
Brief Title: Trial of Tremelimumab in Patients With Previously Treated Metastatic Urothelial Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Matthew Galsky (Other)
Collaborators: AstraZeneca (Industry)
Responsible Party: Sponsor-Investigator, Matthew Galsky, Sponsor-Investigator, Hoosier Cancer Research Network
Organization: Hoosier Cancer Research Network (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HCRN GU17-294
Record Dates: First submitted 2018-06-05; First posted 2018-06-15 (Actual); Results first posted 2024-07-03 (Actual); Last update posted 2024-07-03 (Actual); Status verified 2024-06

CONDITIONS: Urothelial Carcinoma
MeSH Terms: conditions — Carcinoma, Transitional Cell | interventions — tremelimumab

STUDY DESIGN:
Intervention Model Description: Single group assignment
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Tremelimumab (Experimental): Tremelimumab 750 mg IV Day 1 of each 28 day cycle. Up to 7 cycles.
  Interventions: Drug: Tremelimumab

INTERVENTIONS:
Drug: Tremelimumab — Tremelimumab 750 mg IV on Day 1 of each 28 day cycle; up to 7 cycles.
  Subjects that complete all initial 7 cycles but later progress during follow up may receive an additional 7 cycles of tremelimumab providing they meet eligibility criteria.

SUMMARY:
This is a phase II trial designed to estimate the activity of single agent tremelimumab in subjects with metastatic urothelial cancer with disease progression despite prior treatment with PD-1/PD-L1 blockade. The primary endpoint is objective response rate and the study will employ a Simon's 2-stage design.

ELIGIBILITY:
Inclusion Criteria:

* Written informed consent and HIPAA authorization for release of personal health information prior to registration. NOTE: HIPAA authorization may be included in the informed consent or obtained separately.
* ECOG Performance Status of 0 or 1 within 14 days prior to registration.
* Histologically or cytologically documented urothelial cancer. Locally advanced (T4b, any N; or any T, N 2-3) or metastatic disease (M1, Stage IV) (also termed TCC or UCC of the urinary tract; including renal pelvis, ureters, urinary bladder, and urethra). Subjects with mixed histologies are eligible provided that the predominant component is urothelial cancer. Locally advanced bladder cancer must be inoperable on the basis of involvement of pelvic sidewall or adjacent viscera (clinical Stage T4b) or bulky nodal metastasis (N2-N3).
* Representative formalin-fixed paraffin-embedded (FFPE) tumor specimens in paraffin blocks (blocks preferred) or at least 15 unstained slides. If archival tissue is not available and the subject is undergoing a standard of care biopsy, tissue from the biopsy is required to be submitted for correlative analyses. Subjects without adequate baseline tumor tissue may be considered for enrollment on a case by case basis after discussion with the sponsor-investigator.
* Measurable disease according to RECIST 1.1 within 28 days prior to registration. At least 1 lesion, not previously irradiated, that can be accurately measured at baseline as ≥10 mm in the longest diameter (except lymph nodes, which must have short axis ≥15 mm) with computed tomography (CT) (preferred) or magnetic resonance imaging (MRI) scans, preferably with IV contrast, and that is suitable for accurate repeated measurements as per RECIST 1.1 guidelines; lesions in a previously irradiated field can be used as a measurable disease provided that there has been demonstrated progression in the lesion.
* A subject with prior brain metastasis may be considered if they have completed their treatment for brain metastasis at least 4 weeks prior to study registration, have been off of corticosteroids for ≥ 2 weeks, and are asymptomatic
* Subjects must have progressed despite prior treatment with anti-PD-1/PD-L1 antibody therapy. In addition, subjects must meet the following criteria:

  * Subjects must not have progressed within 2 months of starting prior anti-PD-1/PD-L1 antibody therapy.
  * Subjects must have received at least 1 line of prior systemic therapy
  * Must not have experienced a toxicity that led to permanent discontinuation of prior immunotherapy.
  * All AEs while receiving prior immunotherapy must have completely resolved or resolved to baseline prior to screening for this study with the exception of endocrine related AEs that are stable on replacement therapy (e.g., steroids, thyroid hormone) which may be considered eligible but must be discussed with the sponsor-investigator.
  * Must not have experienced a ≥ Grade 3 immune related AE or an immune related neurologic (neuro-muscular) or ocular AE of any grade while receiving prior immunotherapy. NOTE: Subjects with endocrine AE of ≤ Grade 2 are permitted to enroll if they are stably maintained on appropriate replacement therapy and are asymptomatic. Must not have required the use of additional immunosuppression other than corticosteroids for the management of an AE, not have experienced recurrence of an AE if re-challenged, and not currently require maintenance doses of > 10 mg prednisone or equivalent per day.
  * Patients with Gr 3 AST/ALT elevation < 8 fold that resolved with steroids without additional immunosuppression can be included (Patients who experienced Hy's law on PD-1/L1 therapy will be excluded)
* Prior cancer treatment must be completed at least 28 days or 5 half-lives (whichever is shorter) prior to first dose of study drug. Subjects must have recovered from all reversible acute toxic effects of the regimen (other than alopecia) to ≤ Grade 1 or baseline.
* Demonstrate adequate organ function as defined in the table below. All screening labs to be obtained within 14 days prior to registration.
* Absolute Neutrophil Count (ANC) ≥ 1500/mm3
* Hemoglobin (Hgb) ≥ 9 g/dL
* Renal
* Calculated creatinine clearance ≥ 30 cc/min OR
* Creatinine ≤ 1.5
* Bilirubin ≤ 1.5 × upper limit of normal (ULN); This will not apply to
* Aspartate aminotransferase (AST) ≤ 2.5 × ULN (≤ 5 x ULN for subjects with hepatic metastases
* Alanine aminotransferase (ALT) ≤ 2.5 × ULN (≤ 5 x ULN for subjects with hepatic metastases
* Evidence of postmenopausal status or negative urinary or serum pregnancy test for female premenopausal subjects. Women will be considered postmenopausal if they have been amenorrheic for 12 months without an alternative medical cause. The following age-specific requirements apply:
* Females of childbearing potential who are sexually active with a non-sterilized male partner must be willing to abstain from heterosexual activity or to use 1 highly of effective method of contraception from the time of informed consent until 90 days after the last dose of tremelimumab. Non-sterilized male partners of a female patient must use male condom plus spermicide throughout this period. See Table 2 for acceptable contraceptive methods.
* Non-sterilized males who are sexually active with a female partner of childbearing potential must use a male condom plus spermicide from screening through 90 days after receipt of the final dose of tremelimumab. Female partners (of childbearing potential) of male subjects must also use a highly effective method of contraception throughout this period

Exclusion Criteria:

* Pregnant or breastfeeding (NOTE: breast milk cannot be stored for future use while the mother is being treated on study).
* Known additional malignancy that is active and/or progressive requiring treatment. Patients with incidental histologic findings of prostate cancer (tumor/node/metastasis stage of T1a or T1b or prostate-specific antigen <10) who have not received hormonal treatment may be included, pending a discussion with the sponsor-investigator
* Treatment with any investigational drug within 28 days prior to registration.
* Prior treatment with an anti-CTLA-4 antibody
* Any unresolved toxicity National Cancer Institute (NCI) CTCAE Version 4.03 Grade ≥ 2 from previous anticancer therapy with the exception of alopecia, vitiligo, and laboratory values defined in the inclusion criteria.

  * Subjects with Grade ≥ 2 neuropathy will be evaluated on a case-by-case basis after consultation with the Sponsor Investigator
  * Subjects with irreversible toxicity not reasonably expected to be exacerbated by treatment with tremelimumab (e.g., hearing loss) may be included after consultation with the sponsor-investigator
* Any concurrent chemotherapy, investigational product, biologic, or hormonal therapy for cancer treatment. Concurrent use of hormonal therapy for non-cancer related conditions (e.g., hormone replacement therapy) is acceptable. Note: Local treatment of isolated lesions, excluding target lesions, for palliative intent is acceptable (e.g., local surgery or radiotherapy)
* Radiation therapy within 14 days of first dose of study drug
* Major surgical procedure within 28 days prior to first dose of study treatment
* History of allogeneic organ transplantation that requires use of immunosuppressive agents
* Active or prior documented autoimmune of inflammatory disorders (including but not limited to inflammatory bowel disease [eg, colitis or Crohn's disease], diverticulitis [with the exception of diverticulosis], systemic lupus erythematosus, Sarcoidosis syndrome [granulomatosis with polyangiitis], Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc). The following are exceptions to this criterion:

  * Subjects with vitiligo
  * Subjects with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement
  * Any chronic skin condition that does not require systemic therapy
  * Subjects without active disease in the last5 years may be considered for enrollment after discussion with the sponsor-investigator
  * Subjects with celiac disease controlled by diet alone may be considered for enrollment after discussion with the sponsor-investigator
* QT interval corrected for heart rate using Fridericia's formula (QTcF) ≥470 ms calculated. Any clinically significant abnormalities detected require triplicate ECG results and a mean QTcF <470 ms calculated from 3 ECGs obtained over a brief period (eg, 30 minutes)
* Past medical history of Interstitial Lung Disease (ILD), drug-induced ILD, radiation pneumonitis which required steroid treatment, or any evidence of clinically active interstitial lung disease.
* History of active primary immunodeficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2018-11-12 (Actual); Primary Completion 2021-12-06 (Actual); Study Completion 2023-06-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Matthew D Galsky, MD, Principal Investigator — Icahn School of Medicine at Mount Sinai
Locations (7):
- United States (7):
  - Georgetown University, Washington D.C., District of Columbia
  - Winship Cancer Institute of Emory University, Atlanta, Georgia
  - University of Kansas Medical Center Research Institute, Inc., Westwood, Kansas
  - Dana Farber- Partners Cancer Care, Inc, Boston, Massachusetts
  - Ichan School of Medicine at Mount Sinai, New York, New York
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Huntsman Cancer Institute University of Utah, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Miller EJ, Rose TL, Maughan BL, Milowsky MI, Bilen MA, Carthon BC, Gao X, Rapisuwon S, Zhao Q, Yu M, Agarwal N, Galsky MD. Phase 2 trial of tremelimumab in patients with metastatic urothelial cancer previously treated with programmed death 1/programmed death ligand 1 blockade. Cancer. 2024 May 1;130(9):1642-1649. doi: 10.1002/cncr.35179. Epub 2024 Jan 5. PMID 38180804

RESULTS

PARTICIPANT FLOW:
Groups:
- Tremelimumab: Tremelimumab 750 mg IV Day 1 of each 28 day cycle. Up to 7 cycles.
  Tremelimumab: Tremelimumab 750 mg IV on Day 1 of each 28 day cycle; up to 7 cycles.
  Subjects that complete all initial 7 cycles but later progress during follow up may receive an additional 7 cycles of tremelimumab providing they meet eligibility criteria.
Period: Overall Study
Arm/Group | Tremelimumab
Started | 26
Completed | 26
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Tremelimumab
Number analyzed (Participants) | 26
Age, Continuous [Median (Full Range); unit: years] | 71 [48 to 84]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 24
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 5
  White | 19
  More than one race | 0
  Unknown or Not Reported | 1
Region of Enrollment [Number; unit: participants]
  United States | 26
Primary Tumor Site [Count of Participants; unit: Participants]
  Renal Pelvis | 6
  Ureter | 2
  Urinary Bladder | 18

OUTCOME MEASURES:

1. Primary Outcome: Objective Response Rate
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD.
  ORR is defined as the proportion of all subjects with confirmed PR or CR according to RECIST 1.1.
Time Frame: Up to a maximum of 12 months
Population: Out of 26, two patients were not evaluable for response.
Measure: Number; unit: Percentage of participants
Arm/Group | Tremelimumab
Number analyzed (Participants) | 24
Percentage of participants | 8.3

2. Secondary Outcome: Adverse Events
Description: Number of participants with adverse events are reported according to the National Cancer Institute's Common Terminology Criteria for Adverse Events(CTCAE) version 4.
Time Frame: AE had been recorded from time of consent until 30 days after discontinuation of study drug or until a new anti-cancer treatment starts, whichever occurs first; up to a maximum of 13 months
Measure: Count of Participants; unit: Participants
Arm/Group | Tremelimumab
Number analyzed (Participants) | 26
Participants
  Number of patients had at least one grade 3 or greater adverse event | 19
  Number of patients had at least one grade 3 or greater treatment related adverse event | 11
  Number of patients having serious adverse event | 14

3. Secondary Outcome: Disease Control Rate
Description: The disease control rate is defined as the percentage of patients who have achieved complete response, partial response and stable disease by RECIST 1.1
Time Frame: Up to a maximum of 12 months
Population: Out of 26, two patients were not evaluable for response.
Measure: Number; unit: Percentage of participants
Arm/Group | Tremelimumab
Number analyzed (Participants) | 24
Percentage of participants | 29.17

4. Secondary Outcome: Duration of Response
Description: Duration of response (DoR) is defined as the time from randomization to disease progression or death in patients who achieve complete or partial response.
Time Frame: Up to a maximum of 24 months
Population: Out of 26, two patients were not evaluable for response.
Measure: Median (Full Range); unit: Months
Arm/Group | Tremelimumab
Number analyzed (Participants) | 24
Months | 17.45 [10.91 to 23.98]

5. Secondary Outcome: Progression Free Survival (PFS)
Description: Per Response Evaluation Criteria In Solid Tumors Criteria (RECIST): Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Progressive Disease (PD) >= 20% increase in tumor burden relative to nadir or the appearance of one or more new lesions; Stable Disease (SD), not meet criteria for CR/PR/PD.
  PFS is defined as time from registration until disease progression met by RECIST 1.1 or death from any cause.
Time Frame: Time of treatment start until the criteria for disease progression or death. Up to a maximum of 24 months.
Population: Out of 26 patients, only 24 patients were evaluable for PFS.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tremelimumab
Number analyzed (Participants) | 24
Months | 1.83 [1.68 to 1.91]

6. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from treatment start until death or date of last contact.
Time Frame: Time of treatment start until death or date of last contact, up to a maximum of 42 months.
Measure: Median (95% Confidence Interval); unit: Months
Arm/Group | Tremelimumab
Number analyzed (Participants) | 26
Months | 7.75 [5.39 to 15.44]

ADVERSE EVENTS:
Time Frame: All-Cause Mortality was monitored up to a maximum of 42 months. Serious Adverse Events and Other (Not Including Serious) Adverse Events were monitored up to 13 months.
Description: The Adverse Event data reported below reports each CTCAEV4 term individually per each arm/group.
Arm/Group | Tremelimumab
All-Cause Mortality (participants affected / at risk) | 19/26
Serious Adverse Events (participants affected / at risk) | 14/26
Other Adverse Events (participants affected / at risk) | 22/26
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tremelimumab (N=26)
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 3 (3)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 1 (2)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 1 (1)
COLITIS (Gastrointestinal disorders) | 2 (2)
COLONIC OBSTRUCTION (Gastrointestinal disorders) | 1 (1)
CREATININE INCREASED (Investigations) | 2 (2)
DIARRHEA (Gastrointestinal disorders) | 3 (4)
ENCEPHALOPATHY (Nervous system disorders) | 1 (1)
GENERAL DISORDERS AND ADMINISTRATION SITE CONDITIONS - OTHER, SPECIFY (General disorders) | 1 (1)
HEPATIC FAILURE (Hepatobiliary disorders) | 1 (1)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 1 (1)
ILEAL OBSTRUCTION (Gastrointestinal disorders) | 1 (1)
INVESTIGATIONS - OTHER, SPECIFY (Investigations) | 1 (1)
METABOLISM AND NUTRITION DISORDERS - OTHER, SPECIFY (Metabolism and nutrition disorders) | 2 (5)
MULTI-ORGAN FAILURE (General disorders) | 1 (1)
PAIN (General disorders) | 1 (2)
PULMONARY EDEMA (Respiratory, thoracic and mediastinal disorders) | 1 (1)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 1 (2)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SEPSIS (Infections and infestations) | 3 (3)
THROMBOEMBOLIC EVENT (Vascular disorders) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Tremelimumab (N=26)
ADRENAL INSUFFICIENCY (Endocrine disorders) | 2 (2)
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 3 (3)
ALKALINE PHOSPHATASE INCREASED (Investigations) | 6 (7)
ANEMIA (Blood and lymphatic system disorders) | 8 (15)
ANOREXIA (Metabolism and nutrition disorders) | 6 (6)
ANXIETY (Psychiatric disorders) | 2 (2)
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 2 (2)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 3 (4)
BACK PAIN (Musculoskeletal and connective tissue disorders) | 3 (3)
BRUISING (Injury, poisoning and procedural complications) | 1 (1)
CHILLS (General disorders) | 1 (1)
COLITIS (Gastrointestinal disorders) | 2 (3)
CONSTIPATION (Gastrointestinal disorders) | 2 (2)
CREATININE INCREASED (Investigations) | 7 (16)
DELIRIUM (Psychiatric disorders) | 1 (1)
DEPRESSION (Psychiatric disorders) | 1 (1)
DIARRHEA (Gastrointestinal disorders) | 11 (14)
DIZZINESS (Nervous system disorders) | 2 (2)
DRY MOUTH (Gastrointestinal disorders) | 2 (2)
DRY SKIN (Skin and subcutaneous tissue disorders) | 1 (1)
DYSGEUSIA (Nervous system disorders) | 1 (1)
DYSPNEA (Respiratory, thoracic and mediastinal disorders) | 2 (3)
FALL (Injury, poisoning and procedural complications) | 2 (2)
FATIGUE (General disorders) | 12 (14)
FEVER (General disorders) | 2 (2)
GASTROINTESTINAL DISORDERS - OTHER, SPECIFY (Gastrointestinal disorders) | 2 (2)
HEADACHE (Nervous system disorders) | 2 (2)
HEMATURIA (Renal and urinary disorders) | 1 (2)
HOARSENESS (Respiratory, thoracic and mediastinal disorders) | 1 (1)
HOT FLASHES (Vascular disorders) | 1 (1)
HYPERCALCEMIA (Metabolism and nutrition disorders) | 1 (2)
HYPERGLYCEMIA (Metabolism and nutrition disorders) | 3 (9)
HYPERKALEMIA (Metabolism and nutrition disorders) | 4 (5)
HYPERTENSION (Vascular disorders) | 3 (5)
HYPERTHYROIDISM (Endocrine disorders) | 1 (1)
HYPOALBUMINEMIA (Metabolism and nutrition disorders) | 4 (5)
HYPOCALCEMIA (Metabolism and nutrition disorders) | 1 (3)
HYPOGLYCEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPOKALEMIA (Metabolism and nutrition disorders) | 2 (3)
HYPOMAGNESEMIA (Metabolism and nutrition disorders) | 1 (1)
HYPONATREMIA (Metabolism and nutrition disorders) | 9 (14)
HYPOTENSION (Vascular disorders) | 1 (1)
LIPASE INCREASED (Investigations) | 5 (10)
LYMPHOCYTE COUNT DECREASED (Investigations) | 3 (3)
METABOLISM AND NUTRITION DISORDERS - OTHER, SPECIFY (Metabolism and nutrition disorders) | 1 (1)
MUCOSITIS ORAL (Gastrointestinal disorders) | 1 (2)
MUSCLE WEAKNESS LOWER LIMB (Musculoskeletal and connective tissue disorders) | 1 (2)
MUSCULOSKELETAL AND CONNECTIVE TISSUE DISORDER - OTHER, SPECIFY (Musculoskeletal and connective tissue disorders) | 3 (3)
NAUSEA (Gastrointestinal disorders) | 8 (9)
NERVOUS SYSTEM DISORDERS - OTHER, SPECIFY (Nervous system disorders) | 1 (1)
NEUTROPHIL COUNT DECREASED (Investigations) | 1 (1)
PAIN (General disorders) | 1 (2)
PALPITATIONS (Cardiac disorders) | 1 (1)
PAPULOPUSTULAR RASH (Infections and infestations) | 2 (2)
PELVIC PAIN (Reproductive system and breast disorders) | 1 (1)
PLATELET COUNT DECREASED (Investigations) | 3 (3)
PROTEINURIA (Renal and urinary disorders) | 1 (1)
PRURITUS (Skin and subcutaneous tissue disorders) | 5 (5)
RASH ACNEIFORM (Skin and subcutaneous tissue disorders) | 3 (5)
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 4 (4)
RENAL AND URINARY DISORDERS - OTHER, SPECIFY (Renal and urinary disorders) | 1 (1)
RESPIRATORY, THORACIC AND MEDIASTINAL DISORDERS - OTHER, SPECIFY (Respiratory, thoracic and mediastinal disorders) | 1 (1)
SERUM AMYLASE INCREASED (Investigations) | 3 (4)
SINUS TACHYCARDIA (Cardiac disorders) | 1 (1)
SKIN AND SUBCUTANEOUS TISSUE DISORDERS - OTHER, SPECIFY (Skin and subcutaneous tissue disorders) | 1 (1)
THROMBOEMBOLIC EVENT (Vascular disorders) | 1 (1)
URINARY TRACT INFECTION (Infections and infestations) | 3 (3)
URTICARIA (Skin and subcutaneous tissue disorders) | 1 (1)
VOMITING (Gastrointestinal disorders) | 1 (1)
WEIGHT LOSS (Investigations) | 2 (4)
WHITE BLOOD CELL DECREASED (Investigations) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-03-28): https://cdn.clinicaltrials.gov/large-docs/18/NCT03557918/Prot_SAP_000.pdf